CLINICAL TRIAL: NCT03879005
Title: Split Renal Function Using 99mTc-DTPA Versus 99mTc-DMSA in Kidney Patients of Wide Age Ranges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Fathy, Principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SRF using DTPA Vs DMSA
Record Dates: First submitted 2019-03-08; First posted 2019-03-18 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: The Difference in Estimation of Split Renal Function Using the Two Radiopharmaceuticals:Tc-99m DTPA & Tc-99m DMSA in Kidney Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal scintigraphy (Other): 5 mci of 99mTc-DTPA or 99mTc-DMSA is injected once IV. Dose is adjusted according to age and weight.
  Interventions: Other: renal scintigraphy

INTERVENTIONS:
Other: renal scintigraphy — 99mTc-DTPA Scintigraphy Five mci of 99mTc-DTPA will be injected by IV route together with diuretic. Dose will be adjusted according to the age and weight of the patients. A total of 20 min dynamic imaging followed by calculation of GFR and SRF according to the built-in processing protocol Gate's method.
  99mTc-DMSA scintigraphy Five mci of 99mTc- DMSA will be injected by IV route with adjustment according to age and weight. Static images will be acquired in the posterior, anterior, andposterior oblique projections for 60 s each.
  Other Names: 99mTc-DTPA & 99mTc-DMSA renal scintigraphy

SUMMARY:
To evaluate split renal function using Tc-99m DTPA versus Tc-99m DMSA.

DETAILED DESCRIPTION:
Split renal function (SPR) is a determination of the relative contribution of each of the two kidneys . It gives a useful information in several conditions such as evaluating unilateral renal disorders, assessing individual kidney function before and after intervention, and before live donor nephrectomy. Different radiopharmaceuticals such as technetium-99m dimercaptosuccinic acid (99mTc-DMSA), technetium-99m diethylenetriaminepentaaceticacid (99mTc-DTPA), technetium-99m mercaptoacetyltriglycine (99mTc-MAG3), Iodine 131 orthoiodohippurate and more recently technetium-99 m ethylenedicysteine (99mTc-EC) were used, However, 99mTc-DMSA as a static renal agent is considered the most reliable method to measure relative renal function and the most appropriate tracer for renal cortical imaging . In some papers, it is emphasized that relative renal function calculated with 99mTc-DTPA is as reliable as 99mTc-DMSA .‬ The investigators design the study to evaluate the difference in estimation of split renal function using the available two radiopharmaceuticals: Tc-99m DTPA and Tc-99m DMSA.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney patients of wide age ranges.
2. Patients with renal disorders who referred for DMSA and DTPA split renal function.
3. Patients able to sleep in a fixed position for 20 minutes.

Exclusion Criteria:

1. Children unable to sit calm without movement during imaging.
2. Severely ill patients.
3. Patients with allergy to one or more of material method.

Ages: 2 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Split renal function using 99mTc-DTPA versus 99mTc-DMSA in kidney patients of wide age ranges. | one year
  To emphasize that split renal function calculated with Tc-99m DTPA is as reliable as Tc-99m DMSA

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AH Mekkawy, professor, Study Director — Assiut University

REFERENCES:
- [Result] Ardela Diaz E, Miguel Martinez B, Gutierrez Duenas JM, Diez Pascual R, Garcia Arcal D, Dominguez Vallejo FJ. [Comparative study of differential renal function by DMSA and MAG-3 in congenital unilateral uropathies]. Cir Pediatr. 2002 Jul;15(3):118-21. Spanish. PMID 12601986
- [Result] Cao X, Xu X, Grant FD, Treves ST. Estimation of Split Renal Function With 99mTc-DMSA SPECT: Comparison Between 3D Volumetric Assessment and 2D Coronal Projection Imaging. AJR Am J Roentgenol. 2016 Dec;207(6):1324-1328. doi: 10.2214/AJR.16.16307. Epub 2016 Sep 13. PMID 27623376
- [Result] Celik T, Yalcin H, Gunay EC, Ozen A, Ozer C. Comparison of the Relative Renal Function Calculated with 99mTc-Diethylenetriaminepentaacetic Acid and 99mTc-Dimercaptosuccinic Acid in Children. World J Nucl Med. 2014 Sep;13(3):149-53. doi: 10.4103/1450-1147.144812. PMID 25538484
- [Result] Lee WG, Kim JH, Kim JM, Shim KM, Kang SS, Chae HI, Choi SH. Renal uptakes of 99mTc-MAG3, 99mTc-DTPA, and 99mTc-DMSA in rabbits with unilateral ureteral obstruction. In Vivo. 2010 Mar-Apr;24(2):137-9. PMID 20363984